CLINICAL TRIAL: NCT02580591
Title: A Phase III, Randomised, Double Blind, Placebo-controlled, Parallel Group, Efficacy, Safety and Tolerability Trial of Once Daily, Oral Doses of Empagliflozin as Adjunctive to Insulin Therapy Over 26 Weeks in Patients With Type 1 Diabetes Mellitus (EASE-3)
Brief Title: Empagliflozin as Adjunctive to Insulin Therapy Over 26 Weeks in Patients With T1DM (EASE-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.72; 2014-005256-26 (EudraCT Number)
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin

ARMS (4):
- Empagliflozin low dose (Experimental)
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Empagliflozin high dose (Experimental)
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Empagliflozin medium dose (Experimental)
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Arms: Empagliflozin high dose; Empagliflozin low dose; Empagliflozin medium dose
Drug: Placebo — For blinding purposes

SUMMARY:
The study will investigate the efficacy, safety, tolerability and Pharmacokinetic(PK) of 3 doses of empagliflozin compared with placebo over 26 weeks in 960 patients with type 1 diabetes mellitus as adjunctive therapy to insulin

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent
* Male or female patient receiving insulin for the treatment of documented diagnosis of type 1 diabetes mellitus (T1DM) > 1 year
* C-peptide value of < 0.7 ng/mL
* Use of Multiple Daily Injections (MDI) of insulin or insulin pump user with total daily insulin >= 0.3 and <= 1.5 U/kg
* Glycated haemoglobin (HbA1c) >= 7.5% and <= 10.0%
* Good understanding of T1DM
* Age >= 18 years
* Body Mass Index (BMI) >= 18.5 kg/m2
* Estimated glomerular filtration rate >= 30 mL/min/1.73 m2
* Women of child-bearing potential must use highly effective methods of birth control
* Compliance with trial medication administration between 80% and 120% during placebo run-in period Further inclusion criteria apply

Exclusion criteria:

* History of type 2 diabetes mellitus, maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
* Pancreas, pancreatic islet cells or renal transplant recipient
* T1DM treatment with any other antihyperglycaemic drug except subcutaneous basal and bolus insulin within last 3 months
* Occurrence of severe hypoglycaemia within last 3 months and until randomisation
* Occurence of diabetic ketoacidosis within 3 months prior to Visit 1 and until Visit 6
* Irregular sleep/wake cycle
* Acute coronary syndrome, stroke or Transient Ischaemic Attack (TIA) within last 3 months
* Severe gastroparesis
* Brittle diabetes
* Liver disease
* Eating disorders
* Treatment with anti-obesity drugs, weight-loss surgery or aggressive diet regimen
* Treatment with systemic corticosteroids
* Change in dose of thyroid hormones within last 6 weeks and until randomisation
* Cancer or treatment for cancer in the last five years
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells
* Women who are pregnant, nursing, or who plan to become pregnant whilst in the trial
* Alcohol or drug abuse
* Intake of an investigational drug in another trial within last 30 days Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (189):
- United States (39):
  - Healthscan Clinical Trials LLC, Montgomery, Alabama
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Research, Fresno, California
  - Marin Endocrine Care and Research, Greenbrae, California
  - Pacific Research Partners, LLC, Oakland, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - William Sansum Diabetes Center, Santa Barbara, California
  - University of Colorado Denver, Aurora, Colorado
  - International Research Associates, LLC, Hialeah, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Sestron Clinical Research, Marietta, Georgia
  - Eagle's Landing Diabetes and Endocrinology, Stockbridge, Georgia
  - Northwest Endo Diabetes Research, LLC, Arlington Heights, Illinois
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - MODEL Clinical Research, Baltimore, Maryland
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Endocrine-Diabetes Care and Resource Center, Rochester, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Diabetes Endocrinology Research Center of Western New York, Williamsville, New York
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - Holzer Clinic LLC, Gallipolis, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Strand Physician Specialists dba Carolina Health Specialists, Myrtle Beach, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Holston Medical Group, Bristol, Tennessee
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology PA, Austin, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Virginia Endocrinology Research, Chesapeake, Virginia
- Australia (4):
  - Coffs Endocrine & Diabetes Services, Coffs Harbour, New South Wales
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - SA Endocrine Research P/L, Keswick, South Australia
  - Eastern Clinical Research Unit, East Ringwood, Victoria
- Canada (8):
  - Richmond Road and Diagnostic Treatment Centre, Calgary, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Eastern Health (MUN), St. John's, Newfoundland and Labrador
  - Centre for Studies in Family Medicine, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Omnispec Recherche Clinique Inc., Mirabel, Quebec
  - Applied Medical Informatics Research INC., Westmount, Quebec
  - Clinique des maladies Lipidiques de Quebec, Québec
- Czechia (7):
  - University Hospital Brno, Brno
  - Diahaza s.r.o.Intern.Med.Outpat.Clin.Dep.Diabetology,Holesov, Holešov
  - AIDIN VK s.r.o.,Department Diabetology, Hranice, Hranice
  - Univ. Hospital Kralovske Vinohrady, Prague
  - DiaGolfova s.r.o., Department Diabetology, Prague, Prague
  - Milan Kvapil s.r.o.,Diabetology ambulance,Prague, Prague
  - ResTrial s.r.o.Diabetology Ambulance,Prague, Prague
- Finland (5):
  - HUS, Lihavuustutkimusyksikkö Biomedicum Helsinki, Helsinki
  - Mehiläinen Jyväskylä, Jyväskylä
  - Satakunnan Diabetesasema, Pori, Pori
  - FinnMedi Oy, Tampere, Tampere
  - TYKS, Turku
- France (7):
  - HOP Jean Minjoz, Besançon
  - HOP Le Creusot, Le Creusot
  - HOP Paris Saint-Joseph, Paris
  - HOP Bichat, Paris
  - HOP de Poitiers, Poitiers
  - HOP Civil, Strasbourg
  - HOP Rangueil, Toulouse Cédex 04
- Germany (11):
  - Diabetes-Klinik Bad Mergentheim GmbH & Co. KG, Bad Mergentheim
  - Diabetologische Schwerpunktpraxis, Bosenheim, Bosenheim
  - Praxis Dr. Busch, Dortmund, Dortmund
  - GWT-TUD GmbH, Dresden
  - ZKS Südbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Praxis Dr. Kaiser, Frankfurt, Frankfurt
  - Institut für Diabetesforschung Münster GmbH, Münster
  - Diabetologische Schwerpunktpraxis, Münster
  - Praxis Dr. Behnke, Neuwied, Neuwied
  - Praxis Dr. Hilgenberg, Rehburg-Loccum
- Greece (6):
  - "Korgialeneio-Benakeio" Hellenic Red Cross Hospital, Athens
  - General Hospital of Athens "Laiko", Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General Hospital of Nikaia, Nikaia
  - General Hopsital of Thessaloniki "Ippokrateio", Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (7):
  - Clinexpert Kft., Budapest
  - Synexus Magyarorszag Kft., Budapest
  - University Debrecen Hospital, Debrecen
  - CRU Hungary Ltd, Private Practice, Miskolc, Miskolc
  - Clinfan SMO Ltd., Szekszárd
  - Csongrad Country Dr Bugyi Istvan Hosp., Szentes
  - Zala Country Hospital, Diabetic Outpatient Clinic, Zalaegerszeg
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (9):
  - Inrca-Irccs, Ancona
  - A.O. Spedali Civili di Brescia, Brescia
  - Osp. Campo di Marte, Lucca
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Policlinico Gemelli, Roma
  - Osp. S. Giovanni Calibita Fatebenefratelli, Roma
  - IRCCS Gruppo Multimedica, Sesto San Giovanni (MI)
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Ospedale Molinette, AO Città della Salute e della, Torino
- Latvia (7):
  - Zemgales Center of diabetes, Jelgava, Jelgava
  - A. Lucenko's Internist & Endocrinologist Doctor's Practice, Liepāja
  - Dace Teterovska Doctor's Practice in Endocrinology,Ogre, Ogre
  - P. Stradins Clinical University Hospital, Riga, Riga
  - Riga Health Center, Private Practice, Riga
  - Sigulda Hospital, Outpatient department, Sigulda
  - VSV Centrs, Stalte Private Practice, Talsi, Talsi
- Mexico (5):
  - Clínica EndocrInol en Diabetes Obesidad y Tiroides (DOT), Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Unidad de Investigacion Clinica Cardiometabolica de Occident, Guadalajara
  - Instituto Jaliscience de Inv. en Diabetes y Obesidad, S.C., Guadalajara
  - Unidad de Patologia Clinica, Guadalajara
- Netherlands (6):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente locatie Almelo, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - EB Utrecht Research, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (2):
  - South Pacific Clinical Trials, Auckland, New Zealand
  - Lipid and Diabetes Research Group, Christchurch
- Norway (4):
  - M3 Helse AS, Hamar
  - Oslo Universitetssykehus HF, Lipidklinikken, Oslo
  - Stavanger Helseforskning, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (12):
  - DiabSerwis S.C., Chorzow, Chorzów
  - Medical Centre Pratia Gdynia, Gdynia
  - Medical Centre Pratia Katowice I, Katowice
  - Medical Centre Pratia Krakow, Krakow
  - University Hospital in Krakow, Krakow
  - Independent Public Clin.Hosp.no1Lublin,Dep.Internal Diseases, Lublin
  - Witold Chodzko Institute Rural Medic,Dep.Diabetology,Lublin, Lublin
  - Reg.Spec.Hosp.Olsztyn,Clin,Endocrinology,Diabetics.&Int.Med., Olsztyn
  - Clinical Research Center Medicome, Oswiecim, Oświęcim
  - Omedica Medical Centre, Poznan, Poznan
  - Medical Centre Pratia Warszawa, Warsaw
  - NZOZ Med-Art.Specialist Clinics, Zory, Żory
- Portugal (7):
  - Hospital de Braga-Escala Braga, Braga
  - Centro Hospitalar da Cova da Beira Hospital Pêro da Covilhã, Covilha
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - H. Santo António - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar São João,EPE, Porto
  - ULSAM, EPE - Hospital de Santa Luzia, Viana do Castelo
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Romania (5):
  - Nicodiab SRL, Bucharest, Bucharest
  - Milit. Cent. Emerg. Univ. Hosp. Dr. Davila, Met. Dis. Dept., Bucharest
  - SC Medical Centre "Sanatatea Ta" SRL, Bucharest, Bucharest
  - SC Pelican Impex SRL, Cabinet Nr. 201, Diabetes Dept., Oradea, Bihor County
  - Centrul Medical Dr Negrisanu SRL, Timișoara
- Russia (6):
  - City Clinical Hospital no. 67, Moscow, Moscow
  - CJSC"Polyclinic complex",Dep.Endocrinology,St.Petersburg, Saint Petersburg
  - City Outpatient dep.no.107;clinc.pharmacology,st.petersburg, Saint Petersburg
  - Medical Academy named after I. Mechnikov, St. Petersburg, Saint Petersburg
  - City Hospital Saint Elizaveta, Dept. Endocrinology, Saint Petersburg
  - Policlinic No. 1 of Russian Academy of Sciences, St. Petersburg, Saint Petersburg
- South Africa (6):
  - LCS Clinical Research Unit, Bryanston
  - TREAD Research, Cape Town
  - Dr Hilton Kaplan, Cape Town
  - Dr. L. A.Distiller, Johannesburg
  - VX Pharma (Pty) Ltd Pretoria, Pretoria
  - Diabetes Care Centre, Pretoria
- Spain (8):
  - Hospital A Coruña, A Coruña
  - CM Avances Médicos, Granada
  - Hospital de la Inmaculada Concepción, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Endo-Diabesidad-Clínica Durán & Asociados, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
- Sweden (5):
  - Ängelholms Sjukhus, Ängelholm
  - CTC Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karlskoga lasarett, Karlskoga
  - Skånes universitetssjukhus, Lund, Lund
  - S3 Clinical Research Centers, Vällingby
- United Kingdom (12):
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Hull Royal Infirmary, Hull
  - Ipswich Hospital, Ipswich
  - Leicester General Hospital, Leicester
  - Guy's Hospital, London
  - King's College Hospital, London
  - St Mary's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queen's Medical Centre, Nottingham
  - George Eliot Hospital, Nuneaton

REFERENCES:
- [Derived] Song C, Dhaliwal S, Bapat P, Scarr D, Bakhsh A, Budhram D, Verhoeff NJ, Weisman A, Fralick M, Ivers NM, Cherney DZI, Tomlinson G, Lovblom LE, Mumford D, Perkins BA. Point-of-Care Capillary Blood Ketone Measurements and the Prediction of Future Ketoacidosis Risk in Type 1 Diabetes. Diabetes Care. 2023 Nov 1;46(11):1973-1977. doi: 10.2337/dc23-0840. PMID 37616393
- [Derived] Rosenstock J, Marquard J, Laffel LM, Neubacher D, Kaspers S, Cherney DZ, Zinman B, Skyler JS, George J, Soleymanlou N, Perkins BA. Empagliflozin as Adjunctive to Insulin Therapy in Type 1 Diabetes: The EASE Trials. Diabetes Care. 2018 Dec;41(12):2560-2569. doi: 10.2337/dc18-1749. Epub 2018 Oct 4. PMID 30287422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, placebo-controlled, double-blind, parallel-group study compared 3 doses of empagliflozin (2.5 milligram (mg), 10 mg, and 25 mg) with placebo in patients with type 1 diabetes mellitus (T1DM) as adjunctive to optimized insulin therapy.
Pre-assignment Details: 6-Week T1DM therapy (insulin) optimisation period followed by a 2-Week placebo run-in period before randomization. Patients who successfully completed both of the periods were randomized into the 26-Week double-blind treatment period. All treatments were administered in addition to optimized insulin therapy.
Groups:
- Placebo Matching Empagliflozin: Patients administered Placebo matching Empagliflozin film-coated tablet orally once daily in addition as adjunctive to optimized insulin therapy for 26 weeks.
- Empagliflozin 2.5 Milligram (mg): Patients administered Empagliflozin 2.5 mg film-coated tablet orally once daily in addition as adjunctive to optimized insulin therapy for 26 weeks.
- Empagliflozin 10 mg: Patients administered Empagliflozin 10 mg film-coated tablet orally once daily in addition as adjunctive to optimized insulin therapy for 26 weeks.
- Empagliflozin 25 mg: Patients administered Empagliflozin 25 mg film-coated tablet orally once daily in addition as adjunctive to optimized insulin therapy for 26 weeks.
Period: Overall Study
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 242 | 242 | 248 | 245
Treated | 241 | 241 | 248 | 245
Completed | 224 | 232 | 235 | 233
Not Completed | 18 | 10 | 13 | 12
Not completed — Adverse Event | 0 | 1 | 2 | 5
Not completed — Protocol Violation | 3 | 2 | 1 | 1
Not completed — Lost to Follow-up | 5 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 6 | 1 | 2 | 3
Not completed — Not treated | 1 | 1 | 0 | 0
Not completed — Other than specified | 3 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): All patients from the Screened set (SCR) who were randomised to trial medication, regardless of whether any trial medication was taken.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 242 | 242 | 248 | 245 | 977
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: RS
  Years | 42.3 (13.2) | 43.4 (14.3) | 42.3 (13.2) | 44.4 (13.6) | 43.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: RS
  Participants
    Female | 126 | 120 | 132 | 121 | 499
    Male | 116 | 122 | 116 | 124 | 478
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: RS
  Participants
    Hispanic or Latino | 215 | 220 | 233 | 224 | 892
    Not Hispanic or Latino | 27 | 22 | 15 | 21 | 85
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: RS
  Participants
    American Indian or Alaska Native | 7 | 0 | 1 | 5 | 13
    Asian | 2 | 2 | 2 | 5 | 11
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
    Black or African American | 5 | 3 | 10 | 4 | 22
    White | 227 | 234 | 234 | 231 | 926
    More than one race | 0 | 3 | 1 | 0 | 4
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 26 for Full Analysis Set (FAS) (Observed Cases [OC])
Description: Change from baseline in Glycated hemoglobin (HbA1c) for full analysis set (FAS) (observed cases [OC]) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomized trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: Full analysis set (FAS) (observed cases [OC]): Patients in the Treated Set (TS) who had a baseline and at least 1 on-treatment HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 238 | 237 | 244 | 242
Percentage (%) | 0.20 (0.05) | -0.09 (0.05) | -0.25 (0.05) | -0.33 (0.05)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); Model includes baseline HbA1c, baseline Estimated glomerular filtration rate (eGFR) as linear covariates and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline HbA1c by visit interaction as fixed effects. Patient is included as random effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.28, 99% CI 2-sided [-0.46 to -0.11], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; Model includes baseline HbA1c, baseline eGFR as linear covariates and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline HbA1c by visit interaction as fixed effects. Patient is included as random effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.45, 97.5% CI 2-sided [-0.60 to -0.30], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.52, 97.5% CI 2-sided [-0.68 to -0.37], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

2. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 26 for Modified Intention-to-treat Population Set (mITT) (Observed Case (OC) - All Data (AD) (OC-AD))
Description: Change from baseline in Glycated hemoglobin (HbA1c) for modified intention-to-treat population set (mITT) (observed case - all data [OC-AD]) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomized trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: Modified intention-to-treat set (mITT) (observed case - all data [OC-AD]): Patients in the TS who had a baseline and at least 1 post-baseline HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 239 | 239 | 246 | 245
Percentage (%) | 0.21 (0.05) | -0.06 (0.05) | -0.23 (0.05) | -0.30 (0.05)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.40 to -0.14], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Median Difference (Final Values) = -0.44, 97.5% CI 2-sided [-0.59 to -0.28], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.50, 97.5% CI 2-sided [-0.66 to -0.35], Standard Error of Mean 0.07 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

3. Secondary Outcome: Rate Per Patient-year of Investigator-reported Symptomatic Hypoglycemic Adverse Events (AEs) With Confirmed Plasma Glucose (PG)
Description: Rate per patient-year of investigator-reported symptomatic hypoglycemic adverse events (AEs) with confirmed plasma glucose (PG) <54 milligram per deciliter (mg/dL) (<3.0 millimoles per litre (mmol/L)) and/or severe hypoglycemic AEs (i.e. all investigator-reported AEs that had confirmed PG <54 mg/dL [<3.0 mmol/L] with symptoms reported and all severe hypoglycemic events that were confirmed by adjudication) is presented for (i) From week 5 to 26 and (ii) From week 1 to 26. Least squares mean is actually an adjusted event rate. This is key secondary endpoints.
Time Frame: Week 5 to Week 26, Week 1 to Week 26
Population: FAS (OC)
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per patient year
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 235 | 237 | 241 | 237
Events per patient year
  Week 5 to 26 | 6.13 [4.83 to 7.78] | 5.77 [4.53 to 7.34] | 7.37 [5.83 to 9.31] | 6.25 [4.94 to 7.91]
  Week 1 to 26 | 6.62 [5.30 to 8.27] | 6.17 [4.93 to 7.73] | 8.33 [6.70 to 10.37] | 6.96 [5.58 to 8.67]
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); For Week 5 to 26, negative binomial model includes baseline rate of hypoglycemia, baseline HbA1c, and baseline Estimated glomerular filtration rate (eGFR) as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects. Log (time at risk [days]) was used as offset; Test type: Superiority; Negative binomial model; Adjusted Rate Ratio (%) = 0.940, 95% CI 2-sided [0.673 to 1.314] — Empagliflozin 2.5 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2752, Negative binomial model; Adjusted Rate Ratio (%) = 1.202, 97.75% CI 2-sided [0.818 to 1.766] — Empagliflozin 10 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9077, Negative binomial model; Adjusted Rate Ratio (%) = 1.020, 97.75% CI 2-sided [0.693 to 1.501] — Empagliflozin 25 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 4: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); For Week 1 to 26, negative binomial model includes baseline rate of hypoglycemia, baseline HbA1c, and baseline Estimated glomerular filtration rate (eGFR) as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects. Log (time at risk [days]) was used as offset; Test type: Superiority; Negative binomial model; Adjusted Rate Ratio (%) = 0.932, 95% CI 2-sided [0.682 to 1.274]
Statistical Analysis 5: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.1438, Negative binomial model — This is a nominal p-value; Adjusted Rate Ratio (%) = 1.258, 95% CI 2-sided [0.925 to 1.713] — Empagliflozin 10 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 6: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.7543, Negative binomial model — This is a nominal p-value; Adjusted Rate Ratio (%) = 1.051, 95% CI 2-sided [0.771 to 1.433] — Empagliflozin 25 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Change from baseline in body weight is presented With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomized trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 238 | 237 | 243 | 240
Kilogram (kg) | 0.21 (0.20) | -1.55 (0.20) | -2.83 (0.20) | -3.22 (0.20)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); Model includes baseline weight, baseline Estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline weight by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.32 to -1.20] — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -3.04, 99.75% CI 2-sided [-3.91 to -2.18] — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -3.43, 99.75% CI 2-sided [-4.30 to -2.57] — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

5. Secondary Outcome: Change From Baseline in Total Daily Insulin Dose (TDID) at Week 26
Description: Change from baseline in Total daily insulin dose (TDID) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomized trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Unit/kilogram (U/kg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 217 | 223 | 217 | 220
Unit/kilogram (U/kg) | -0.011 (0.007) | -0.060 (0.007) | -0.080 (0.007) | -0.102 (0.007)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); Model includes baseline total daily insulin dose, baseline estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline total daily insulin dose by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.069 to -0.030] — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.070, 99.75% CI 2-sided [-0.101 to -0.039] — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.091, 99.75% CI 2-sided [-0.122 to -0.060], Standard Error of Mean 0.010 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 26
Description: Change from baseline in Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomized trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS observed cases excluding data after change in use of anti-hypertensives (OC-H)
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 237 | 236 | 240 | 238
Millimeters of mercury (mmHg)
  SBP | 0.4 (0.7) | -1.7 (0.7) | -3.5 (0.7) | -3.4 (0.7)
  DBP | 0.0 (0.4) | -0.4 (0.4) | -1.8 (0.4) | -1.5 (0.4)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); For SBP, the model includes baseline SBP seated, baseline Estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline SBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; Mixed effect Model Repeat MeasurementMix; Median Difference (Final Values) = -2.1, 95% CI 2-sided [-3.9 to -0.2] — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For SBP, the model includes baseline SBP seated, baseline Estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, , treatment by visit interaction, baseline SBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -3.9, 99.75% CI 2-sided [-6.8 to -1.1] — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -3.7, 99.75% CI 2-sided [-6.6 to -0.9] — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 4: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 2.5 Milligram (mg); For DBP, the model includes baseline DBP seated, baseline Estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline DBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.5 to 0.9] — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 5: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For DBP, the model includes baseline DBP seated, baseline Estimated glomerular filtration rate (eGFR), baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, ß, treatment by visit interaction, baseline DBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0047, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -1.7, 99.75% CI 2-sided [-3.6 to 0.1] — Mean Difference= Empagliflozin 2.5 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 6: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.0202, Mixed effect Model Repeat Measurement; Mean Difference (Final Values) = -1.4, 99.75% CI 2-sided [-3.3 to 0.4]

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication until 7 days after last in-take of trial medication, up to 232 days.
Description: Treated set (TS): All patients who were treated with at least one dose of randomised trial medication, the TS was the basis for safety analyses. The Total Number of Participants at Risk is based on Treated set.
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 2.5 Milligram (mg) | Empagliflozin 10 mg | Empagliflozin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/241 | 0/248 | 1/245
Serious Adverse Events (participants affected / at risk) | 16/241 | 13/241 | 21/248 | 16/245
Other Adverse Events (participants affected / at risk) | 153/241 | 146/241 | 172/248 | 162/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Empagliflozin (N=241) | Empagliflozin 2.5 Milligram (mg) (N=241) | Empagliflozin 10 mg (N=248) | Empagliflozin 25 mg (N=245)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinopathy haemorrhagic (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anion gap increased (Investigations) | 0 | 0 | 1 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 1 | 0
Blood gases abnormal (Investigations) | 0 | 0 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Blood ketone body increased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1 | 0
Acetonaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2 | 6 | 5
Diabetic ketosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 3 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2
Ketosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Vaginal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Empagliflozin (N=241) | Empagliflozin 2.5 Milligram (mg) (N=241) | Empagliflozin 10 mg (N=248) | Empagliflozin 25 mg (N=245)
Nasopharyngitis (Infections and infestations) | 24 | 23 | 22 | 26
Urinary tract infection (Infections and infestations) | 12 | 12 | 9 | 16
Blood ketone body increased (Investigations) | 3 | 4 | 15 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 144 | 137 | 162 | 151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT02580591/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT02580591/SAP_001.pdf